CLINICAL TRIAL: NCT04597970
Title: A Phase II Clinical Study of Transarterial Chemoembolization (TACE) Plus Hepatic Arterial Infusion Chemotherapy (HAIC) With Oxaliplatin and Raltitrexed for Barcelona Stage C Hepatocellular Carcinoma (HCC)
Brief Title: TACE Plus HAIC With Oxaliplatin and Raltitrexed for BCLC Stage C HCC
Acronym: OXRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhu Xu, Hospital Chief Physician，MD, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020YJZ41
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Transarterial Chemoembolization; Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transcatheter arterial chemoembolization; Hepatic arterial infusion chemotherapy; Oxaliplatin; Raltitrexed
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cTACE-HAIC(oxaliplatin and raltitrexed) (Experimental): Patients receive cTACE+HAIC (oxaliplatin, raltitrexed) treatment, 6-8 weeks as a cycle
  Interventions: Drug: cTACE-HAIC

INTERVENTIONS:
Drug: cTACE-HAIC — transarterial chemoembolization (TACE) plus Hepatic Arterial Infusion Chemotherapy (HAIC) with oxaliplatin and raltitrexed for Barcelona stage C hepatocellular carcinoma (HCC)
  Other Names: OXRI

SUMMARY:
Purpose：explore the effectiveness and safety of transarterial chemoembolization (TACE) plus Hepatic Arterial Infusion Chemotherapy (HAIC) with oxaliplatin and raltitrexed for Barcelona stage C hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Thhis is a non-randomized, open, single-arm clinical study. patients receive cTACE+HAIC (oxaliplatin, raltitrexed) treatment, 6-8 weeks as a cycle, until the disease progresses, intolerable toxicity occurs, the patient is lost to follow-up or death, or situations other judged by researchers which treatment should be stopped.

Number of patients: 66 patients End points：primary end points：safety 、objective response rate，disease control rate，progression free overall survival，second end point ：overall survival Include criteria：

1. Volunteer to participate and sign the informed consent in writing;
2. Age: 18-75 years old;
3. No gender limit;
4. BCLC stage C hepatocellular carcinoma with pathological diagnosis or clinical diagnosis;
5. Barcelona stage C patients who failed first-line treatment (including but not limited to sorafenib, levatinib, atelizumab combined with bevacizumab, etc.); they have not received sorafenib in the past The patients treated by Sorafenib can receive sorafenib treatment at the same time, and the patients who have received sorafenib treatment progress can also receive regorafenib treatment.
6. At least one measurable lesion (according to mRECIST criteria) imaging diagnosis time ≤ 21 days from selection;
7. Child-pugh grade A-B7 grade
8. The expected survival period is ≥3 months;
9. ECOG Performance Status (ECOG) 0-2;
10. Sufficient bone marrow hematopoietic function (within 7 days): hemoglobin ≥9 g/dL, white blood cells ≥3.0×109/L, neutrophils ≥1.5x109/L, platelets ≥80x109/L; liver and kidney functions are normal (Within 14 days): TBIL≤1.5 times the upper limit of normal; ALT and AST≤5 times the upper limit of normal; creatinine≤1.5 times the upper limit of normal; INR<1.7 or prolonged PT<4s

Exclude criteria:

1. Those who are currently receiving other effective treatments;
2. Patients who have received oxaliplatin and raltitrexed in the past;
3. Patients who have participated in other clinical trials within 4 weeks before enrollment;
4. Unable to cooperate with cTACE and HAIC treatment;
5. Patients with primary malignant tumors other than hepatocellular carcinoma at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
6. Clinically significant cardiovascular diseases, such as heart failure (NYHA III-IV), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or a history of myocardial infarction within the past 1 year;
7. Neurological or mental abnormalities that affect cognitive ability, including central nervous system transfer;
8. There were active serious clinical infections (>grade 2 NCI-CTCAE version 4.0), including active tuberculosis within 14 days before enrollment;
9. Known or self-reported HIV infection;
10. Uncontrolled systemic diseases, such as poorly controlled diabetes;
11. Known to have hypersensitivity or allergic reactions to any component of the study drug;
12. Pregnancy (determined by serum β-chorionic gonadotropin test) or breast-feeding Treatment：patients receive cTACE+HAIC (oxaliplatin, raltitrexed) treatment, 6-8 weeks as a cycle, until the disease progresses, intolerable toxicity occurs, the patient is lost to follow-up or death, or situations other judged by researchers which treatment should be stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent in writing;
2. Age: 18-75 years old;
3. No gender limit;
4. BCLC stage C hepatocellular carcinoma with clear pathological diagnosis or clinical diagnosis;
5. Barcelona stage C patients who failed first-line treatment (including but not limited to sorafenib, levatinib, atelizumab combined with bevacizumab, etc.); they have not received sorafenib in the past The patients treated by Sorafenib can receive sorafenib treatment at the same time, and the patients who have received sorafenib treatment progress can also receive regorafenib treatment.
6. At least one measurable lesion (according to mRECIST criteria) imaging diagnosis time ≤ 21 days from selection;
7. Child-pugh grade A-B7 grade
8. The expected survival period is ≥3 months;
9. General physical condition (ECOG) 0-2;
10. Sufficient bone marrow hematopoietic function (within 7 days): hemoglobin ≥9 g/dL, white blood cells ≥3.0×109/L, neutrophils ≥1.5x 109/L, platelets ≥80x 109/L; liver and kidney functions are normal (Within 14 days): TBIL≤1.5 times the upper limit of normal; ALT and AST≤5 times the upper limit of normal; creatinine≤1.5 times the upper limit of normal; INR<1.7 or prolonged PT<4s

Exclusion Criteria:

1. Those who are currently receiving other effective treatments;
2. Patients who have received oxaliplatin and raltitrexed in the past;
3. Patients who have participated in other clinical trials within 4 weeks before enrollment;
4. Unable to cooperate with cTACE and HAIC treatment;
5. Patients with primary malignant tumors other than hepatocellular carcinoma at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
6. Clinically significant cardiovascular diseases, such as heart failure (NYHA III-IV), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or a history of myocardial infarction within the past 1 year;
7. Neurological or mental abnormalities that affect cognitive ability, including central nervous system transfer;
8. There were active serious clinical infections (>grade 2 NCI-CTCAE version 4.0), including active tuberculosis within 14 days before enrollment;
9. Known or self-reported HIV infection;
10. Uncontrolled systemic diseases, such as poorly controlled diabetes;
11. Known to have hypersensitivity or allergic reactions to any component of the study drug;
12. Pregnancy (determined by serum β-chorionic gonadotropin test) or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2021-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 6 months
  The objective response rate (ORR) was defined as the complete response (CR) rate + the partial response (PR) rate
Disease control rate, DCR | 6 months
  disease control rate (DCR) was defined as the CR rate + the PR rate + the stable disease (SD) rate
Progression free overall survival，PFS | 8 months
  PFS was defined as the interval between the time at which treatment was initiated and intrahepatic tumor and/or extrahepatic tumor progression, symptomatic progression, including massive ascites and liver function that was categorized as Child-Pugh grade C, or death from any cause

SECONDARY OUTCOMES:
Overall survival， OS | 25 months
  overall survival (OS) was defined as the interval between the time at which treatment was initiated and death or the last follow-up assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhu, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No